CLINICAL TRIAL: NCT00575575
Title: the Research on Suicidal Ideation of University Students in Harbin City and Intervention on Them
Brief Title: Research on Suicidal Ideation of University Students in Harbin City and Cognitive Behavior Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Baofeng Yang, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 196781; 19678181
Record Dates: First submitted 2007-12-15; First posted 2007-12-18 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Suicide
Keywords: Suicidal ideation; cognitive behavior therapy
MeSH Terms: conditions — Suicide; Suicidal Ideation | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A,2 (Experimental)
  Interventions: Behavioral: cognitive behavior therapy

INTERVENTIONS:
Behavioral: cognitive behavior therapy — cognitive behavior therapy once a week

SUMMARY:
The purposes of this research are:

* to understand the status of suicidal ideation, suicidal behavior, and depression in Harbin University students; and
* to analyse the infect factors of suicidal ideation and suicidal behavior.

With cognitive behavior interventions on students with suicidal ideation, suicidal behavior, and middle or high degree of depression, the researchers can provide a scientific and effective intervention to the students.

Cognitive therapy for the prevention of suicide attempts: a randomized controlled trial.

Brown GK, Ten Have T, Henriques GR, Xie SX, Hollander JE, Beck AT. Department of Psychiatry, University of Pennsylvania, Philadelphia 19104, USA. gregbrow@mail.med.upenn.edu JAMA. 2005 Aug 3;294(5):563-70.

DETAILED DESCRIPTION:
By using suicidal ideation scale, to assess the status of suicidal ideation and suicidal attempt in 6000 university students in Harbin city. About 300 students with suicidal ideation and depression disorder randomized into two groups (control and intervention groups) accept the cognitive behavior intervention. We will assess the depression after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Suicidal ideation or the scores of Beck Depression Inventory ≧14

Exclusion Criteria:

* have no Suicidal ideation and the scores of Beck Depression Inventory <14

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 355 (Actual)
Dates: Start 2007-06; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
suicidal ideation; depression | half a year

CONTACTS AND LOCATIONS:
Overall Officials: Yanjie Yang, doctor, Study Director — Harbin Medical University